CLINICAL TRIAL: NCT01191489
Title: Comparison Between High-flow Conditioned Oxygen Therapy and Non-invasive Ventilation in Prevention of Post-extubation Respiratory Failure. A Randomized Controlled Trial
Brief Title: High-flow Conditioned Oxygen Therapy Versus Non-invasive Ventilation: Prevention of Post-extubation Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Infanta Sofia (Other)
Responsible Party: Principal Investigator, Gonzalo Hernandez Martinez, Gonzalo Hernandez Martinez, Hospital Infanta Sofia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HULP-3116
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Post-extubation Respiratory Failure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Flow Conditioned Oxygen Therapy in high risk patients (Experimental)
  Interventions: Device: High Flow Conditioned Oxygen Therapy in High Risk Patients
- Non-invasive mechanical ventilation in High Risk Patients (Active Comparator)
  Interventions: Device: Non-invasive mechanical ventilation
- High Flow Conditioned Oxygen Therapy in Low Risk Patients (Experimental)
  Interventions: Device: High Flow Conditioned Oxygen Therapy in High Risk Patients
- Conventional Oxygen Therapy in Low Risk Patients (Active Comparator)
  Interventions: Device: Conventional Oxygen Therapy

INTERVENTIONS:
Device: High Flow Conditioned Oxygen Therapy in High Risk Patients — OptiFlow system (R) with nasal cannula.
  Arms: High Flow Conditioned Oxygen Therapy in Low Risk Patients; High Flow Conditioned Oxygen Therapy in high risk patients
Device: Non-invasive mechanical ventilation — Bilevel pressure support through a facial mask
  Arms: Non-invasive mechanical ventilation in High Risk Patients
Device: Conventional Oxygen Therapy — Conventional Oxygen Therapy with nasal cannula or Venturi facial mask.
  Arms: Conventional Oxygen Therapy in Low Risk Patients

SUMMARY:
The main aim is to demonstrate whether the high flow conditioned oxygen therapy reduces the reintubation rate. Post-extubation respiratory failure risk will be stratified (as the randomization). In high risk patients high flow conditioned oxygen therapy will be compared with with not conditioned non-invasive mechanical ventilation. In low risk patients comparison will be conventional oxygen therapy. Hypercapnic patients will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Low Risk Patients:
* Any extubated patients after tolerating a spontaneous breathing trial.
* High Risk Patients:
* Any extubated patients after >48 hours under mechanical ventilation and any of the following:
* >65 years

  * cardiac failure as the primary indication of mechanical ventilation
  * COPD
  * APACHE II >12 points the extubation day
  * BMI >30
  * inability to manage respiratory secretions

    * 1 failed spontaneous breathing trial
    * 1 comorbidity
    * 7 days under mechanical ventilation

Exclusion Criteria:

* <18 years
* thacheotomized patients
* recent facial or cervical trauma/surgery
* active gastro-intestinal bleeding
* lack of cooperation and patients with any failed spontaneous breathing trial because of hypercapnia development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Post-extubation respiratory failure and Reintubation rate | 3 months

SECONDARY OUTCOMES:
Intensive Care Unit mortality rate | 3 month
Hospital mortality rate | 6 months
Intensive Care Unit length of stay | 3 months
Hospital length of stay | 6 months
Nosocomial pneumonia rate | 3 months
Tracheobronchitis rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Hernandez, MD, Study Chair — Hospital Infanta Sofia
Locations (2):
- Spain (2):
  - Hospital General de Ciudad Real, Ciudad Real, Ciudad Real
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid

REFERENCES:
- [Derived] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Derived] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498